CLINICAL TRIAL: NCT02045381
Title: Optimization of MRI for Radiation Therapy
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2012.113; HUM00068061 (Other: University of Michigan)
Record Dates: First submitted 2013-12-18; First posted 2014-01-24 (Estimated); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Cancer Liver; Cancer Brain; Cancer Head &Neck; Cancer Pelvis
Keywords: Cancer; MRI
MeSH Terms: conditions — Carcinoma, Hepatocellular; Brain Neoplasms; Head and Neck Neoplasms; Pelvic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MRI group: Patient receives one research MRI prior to radiation treatment.
  Interventions: Procedure: MRI Group

INTERVENTIONS:
Procedure: MRI Group — A single research MRI

SUMMARY:
Currently, appropriate patients undergo MRI imaging with immobilization and sequences optimized for diagnostic radiology purposes. Using a mutual information algorithm, these images are then registered to a treatment planning CT obtained with custom immobilization to minimize intra-and inter-treatment motion and positional variation. This image registration process is time-consuming and introduces additional layers of geometric uncertainty into what should be a highly precise treatment planning process. However, it is necessary, since radiation dose calculations cannot be performed on MRI data due to the lack of crucial density information. The investigator envisions CT-less treatment planning, using only MRI, due to superior imaging characteristics, fully integrated into the radiation oncology clinic. This study will begin this process.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* A working diagnosis of malignancy in the liver, brain, H&N, or pelvis
* A plan to treat with radiotherapy

Exclusion Criteria:

* Patients with contraindications to having a contrast enhanced MRI scan. These contraindications will be assessed at the time of enrollment using the guidelines set up and in clinical use by the Radiology Department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants having a working diagnosis of malignancy in the liver, brain, head and neck, or pelvis, and a plan to treat with radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-03-14 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with MRI images suitable for analyses | Day One
  Patients will be off protocol immediately after the single MRI scan. Comparative treatment planning will occur off-line and will not be used for patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Jolly, MD, Principal Investigator — University of Michigan
Locations (1):
- Univeristy of Michigan, Ann Arbor, Michigan, United States